CLINICAL TRIAL: NCT04424706
Title: The Effect and Mechanism of MMP-9 in Inducing Atherosclerosis in Type 2 Diabetes
Brief Title: The Effect and Mechanism of MMP-9 in Inducing Atherosclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Majianhua (Other)
Responsible Party: Sponsor-Investigator, Majianhua, Head of Department of Endocrinology, Nanjing First Hospital, Nanjing Medical University
Organization: Nanjing First Hospital, Nanjing Medical University (Other)
Other Study IDs: KY20200320-01
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum for testing the MMP-9 level
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal people: No diabetes and atherosclerosis
  Interventions: Diagnostic Test: people without type 2 diabetes or atherosclerosis
- type 2 diabetes mellitus without atherosclerosis: Newly diagnosed type 2 diabetes without atherosclerosis
  Interventions: Diagnostic Test: diagnosed as type 2 diabetes without atherosclerosis
- type 2 diabetes mellitus with atherosclerosis: Newly diagnosed type 2 diabetes with atherosclerosis
  Interventions: Diagnostic Test: diagnosed as type 2 diabetes with atherosclerosis

INTERVENTIONS:
Diagnostic Test: diagnosed as type 2 diabetes without atherosclerosis — patients diagnosed as type 2 diabetes without atherosclerosis
  Groups: type 2 diabetes mellitus without atherosclerosis
Diagnostic Test: diagnosed as type 2 diabetes with atherosclerosis — patients diagnosed as type 2 diabetes with atherosclerosis
  Groups: type 2 diabetes mellitus with atherosclerosis
Diagnostic Test: people without type 2 diabetes or atherosclerosis — normal people without type 2 diabetes or atherosclerosis
  Groups: Normal people

SUMMARY:
The study will assess the serum expression of MMP-9 in normal people, type 2 diabetic patients and type 2 diabetic patients with atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* volunteer to participate and be able to sign informed consent prior to the trial.
* patients with type 2 diabetes, aged 18-60 years old, meeting WHO1999 diagnostic criteria, have not used any drugs.
* The patients have completed carotid ultrasound during hospitalization.

Exclusion Criteria:

* patients with any antidiabetic drugs.
* impaired liver and kidney function with ALT 2.5 times higher than the upper limit of normal value; Serum creatinine was 1.3 times higher than the upper limit of normal.
* drug abuse and alcohol dependence in the past 5 years.
* systemic hormone therapy was used in the last three months.
* patients with infection and stress within 4 weeks.
* any other obvious conditions or associated diseases determined by the researcher: such as severe cardiopulmonary diseases, endocrine diseases, neurological diseases, tumors and other diseases, other pancreatic diseases, history of mental diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal control group, newly diagnosis of type 2 diabetes mellitus with atherosclerosis, newly diagnosis of type 2 diabetes mellitus without atherosclerosis
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
total MMP-9 levels | 6 months
  the different group of total MMP-9 levels

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu B, Su L, Loo SJ, Gao Y, Khin E, Kong X, Dalan R, Su X, Lee KO, Ma J, Ye L. Matrix metallopeptidase 9 contributes to the beginning of plaque and is a potential biomarker for the early identification of atherosclerosis in asymptomatic patients with diabetes. Front Endocrinol (Lausanne). 2024 Apr 10;15:1369369. doi: 10.3389/fendo.2024.1369369. eCollection 2024. PMID 38660518